CLINICAL TRIAL: NCT04347499
Title: The Effect Of Culturally Adapted Cognitive Behaviour Therapy (CaCBT) Based Guided Self-Help in Patients With Postnatal Depression: A Randomised Controlled Trial
Brief Title: Culturally Adapted CBT Based Guided Self-Help in Patients With Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peshawar Medical College (Other)
Collaborators: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Principal Investigator, Muhammad Irfan, Prof. of Psychiatry & Director Research, Peshawar Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT PND KHI
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Postnatal Depression
Keywords: Cognitive Behaviour Therapy; Postnatal Depression; Guided Self Help
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive CaCBT based guided selfhelp using the manual (Khushi Aur Khatoon) as an intervention in addition to treatment as usual
  Interventions: Other: CaCBT based guided self help using Khushi aur Khatoon Manual
- Control (No Intervention): This group will receive treatment as usual

INTERVENTIONS:
Other: CaCBT based guided self help using Khushi aur Khatoon Manual — CaCBT based guided self help using the manual named Khushi Aur Khatoon in the intervention arm
  Arms: Intervention

SUMMARY:
This is a randomized controlled assessor-blind clinical trial comparing CaCBT based guided self-help (using a manual titled Khushi Aur Khatoon) against treatment as usual (TAU)

DETAILED DESCRIPTION:
The prevalence of postnatal depression(PND) in Asian countries ranges from 3.5% to 63.3% where Malaysia and Pakistan have the lowest and highest, respectively. Risk factors for postnatal depression have been clustered into biological/ physical (e.g., Vitamin B Deficiency), psychological (e.g., antenatal depression), obstetric/pediatric (e.g., unwanted pregnancy), socio-demographic (e.g., poverty), and cultural factors (e.g., preference of infants' gender).

Cognitive behaviour therapy (CBT) is the best-studied form of psychotherapy in patients who have had Postnatal Depression, in reducing depressive symptoms. This study is planned to explore the effect of culturally adapted Cognitive Behaviour Therapy (CaCBT) based Guided self-help (using the book, Khushi Aur Khatoon) compared with treatment as usual in improving depression in PND patients. Participants visiting a tertiary care hospital in Karachi, who meet the entry criteria will be randomly allocated to one of the groups, i.e., CaCBT (Intervention group) or TAU (Control Group) in a 1:1 ratio. after taking written informed consent.

The sample size calculation is based on the assumption of using an Analysis of Covariance (ANCOVA) to analyze the outcome while controlling for baseline and is based on formulas given by Van Breukelen GJP and Borm GF et al. The investigators assume a correlation between baseline EPDS and endpoint EPDS of 0.5, 90% power, and a significance level of 0.05 with the two-sided test. A sample of 48 subjects per group is sufficient to achieve the expected power to detect an effect size equivalent to Cohen's d=0.3, which is a small to medium effect size. Considering means and standard deviations, this effect is equivalent to a difference of 0.8 points at the post, between the groups, in average EPDS score. To accommodate for up to 30% of dropouts, the investigators plan to recruit 140 participants in the study.

Participants were assessed at baseline and 9-12 weeks (end of therapy) from baseline. The primary outcome measure was the Edinburgh Postnatal Depression Scale (EPDS). The secondary outcome measures include Bradford Somatic Inventory (BSI) and World Health Organization Disability Assessment Schedule (WHO DAS 2.0). The investigators also measured satisfaction with the treatment at the end of therapy using a visual analog scale from the intervention group.

The investigators followed the CONSORT guidelines for reporting randomized controlled trials. The analyses were carried out on an intention-to-treat basis using SPSS version 25. Comparisons for intention-to-treat analysis participants were included in the groups to which they are randomized regardless of how long or even whether they received the treatment allocated to them or not. Missing values were imputed using the last observation carried forward (LOCF) method. Both Chi-Square and t-tests were used for baseline comparisons. End-of-therapy scores on various outcome measures between the Intervention and the Control groups were compared using an Analysis of Covariance (ANCOVA) to adjust for baseline scores.

ELIGIBILITY:
Inclusion Criteria:

* Score of 10 or more on EPDS
* Fulfilling criteria of Major Depressive Disorder using DSM-V with a specifier of Peripartum Onset.

Exclusion Criteria:

* Participants with use of alcohol or drugs
* Significant cognitive impairment (intellectual disability or dementia)
* Active psychosis
* Participants who have received CBT during the previous 12 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 9-12 weeks (end of therapy)
  Change in the score of Edinburgh Postnatal Depression (EPDS) from baseline to end of therapy Minimum Score = 0 Maximum Score = 30 Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder.
  Higher scores means a worse outcome.

SECONDARY OUTCOMES:
Bradford Somatic Inventory (BSI) | 9-12 weeks (end of therapy)
  Change in the score of Bradford Somatic Inventory (BSI) from baseline to end of therapy Minimum Score = 0 Maximum Score = 92 Higher scores mean a worse outcome.
World Health Organisation Disability Assessment Schedule (WHODAS 2.0) | 9-12 weeks (end of therapy)
  Change in the score of World Health Organisation Disability Assessment Schedule (WHODAS 2.0) from baseline to end of therapy Minimum Score = 0 Maximum Score = 48 Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, PhD, Study Chair — University of Toronto
Locations (1):
- Zainab Panjwani Hospital, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No